CLINICAL TRIAL: NCT03815604
Title: Independent Housing and Support for People With Severe Mental Illness: Randomized Controlled Trial vs. Observational Study
Brief Title: Independent Housing and Support for People With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Zurich (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10531C_179451
Record Dates: First submitted 2018-12-04; First posted 2019-01-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Severe Mental Disorder
Keywords: Psychiatric Rehabilitation; Supported Housing; Residential Care
MeSH Terms: conditions — Mental Disorders | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: As the preference issue makes RCTs in housing research difficult the investigators will use a specific time window in Zurich that allows conducting an RCT due to a scarcity of IHS settings and will combine the RCT with a comparative observational study in Berne where IHS is already well-established.
  The investigators intend to directly compare the outcomes of a randomized controlled trial (RCT) with a study in an observational study design (OSD). Here, the investigators utilize the hypothesis that the OSD will provide similar results as the RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RCT-IHS (Experimental): Behavioral: At the Zurich site, the experimental intervention is called Independent Housing and Support
  Interventions: Behavioral: Independent Housing and Support (IHS)
- RCT-RCS/TAU (Active Comparator): Behavioral: At the Zurich site, the comparator is usual residential care
  Interventions: Behavioral: Residential Care Settings and other Treatment as Usual (RCS/TAU)
- OSD-IHS (Experimental): Behavioral: At the Berne site, the experimental intervention is called Independent Housing and Support
  Interventions: Behavioral: Independent Housing and Support (IHS)
- OSD-RCS/TAU (Active Comparator): Behavioral: At the Berne site, the comparator is usual residential care
  Interventions: Behavioral: Residential Care Settings and other Treatment as Usual (RCS/TAU)

INTERVENTIONS:
Behavioral: Independent Housing and Support (IHS) — Direct placement of people with SMI in an independent accommodation in the community, usually in a flat rented by the service user. Support is provided by a coach according to individual needs in a permanent housing situation without time limit.
  Arms: OSD-IHS; RCT-IHS
Behavioral: Residential Care Settings and other Treatment as Usual (RCS/TAU) — Placement in a common residential home or supportive housing setting with the aim to gain psycho-social stability before being able to maintain independent housing.
  Arms: OSD-RCS/TAU; RCT-RCS/TAU

SUMMARY:
Background: Adequate and stable housing conditions are fundamental for the psychiatric rehabilitation of individuals with severe mental illness (SMI). A common approach in psychiatric rehabilitation relies on a continuum of residential services that aims at enabling the person with SMI to live eventually independently. Current state of research, however, shows clearly that most persons in question remain in residential care settings or other treatment as usual conditions (RCS/TAU). The Independent Housing and Support (IHS) scheme is a new model that aims at direct placement in an independent accommodation in the community. Support is provided according to individual needs in a permanent housing situation without time limit. Up to now, randomized controlled trials (RCTs) to evaluate the effectiveness of IHS have only been conducted with homeless populations in North America. The purpose of the present study is to evaluate IHS compared to traditional RCS/TAU for non-homeless persons with severe mental illness. With this study, the investigators aim at demonstrating that IHS is not inferior to RCS/TAU. The rationale for utilizing a non-inferiority approach is based on the current state of research and on research that has shown strong preferences for IHS against RCS/TAU by people with SMI.

Methods: As the preference issue makes RCTs in housing research difficult the investigators will use a specific time window in Zurich that allows conducting a RCT due to a scarcity of IHS settings and will combine the RCT with a comparative observational study in Berne where IHS is already well-established. At the Zurich site, a RCT compares the effects of living with IHS against living in residential care. At the Berne site, an observational study design (OSD) will be applied in connection with the same types of housing as in Zurich. Propensity scoring will be utilized to minimize the risk of bias in the OSD. A number of N=56 eligible subjects in Zurich and N=112 subjects (due to specific requirements for propensity scoring) in Berne complying with the inclusion criteria will be recruited and allocated to intervention and control groups according to the site-specific study designs. Recruitment period will last 21 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary mental disorder according to ICD-10-categories
* Age 18 to 65 years
* Ability to communicate in German language
* Ability to give informed consent
* Written informed consent as documented by signature
* Ability to take medication if indicated
* Willingness to handle out of pocket expenses or established assistance by custodian/guardian

Exclusion Criteria:

* Severe learning disability, intoxication, delirium, dementia
* Participants lacking capacity
* Indication for hospital treatment due to acute symptomatology at admission
* Acute endangerment of self or others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Social Functioning Scale (SFS) | Change from baseline (T0) to 24 months (T3)
  The SFS is a self-rating questionnaire and will be used to assess changes in participant's social inclusion in terms of the following subscales: 1) social engagement/withdrawal, 2) interpersonal behavior, 3) independence-performance, 4) independence-competence, 5) recreation, 6) pro-social activities, and 7) employment/occupation. The SFS includes 76 items in a varying answer format. In 68 items, participants are asked to answer on a 4-point Likert scale. The total-score ranges from 0 to 135 with higher score indicating better social inclusion.

SECONDARY OUTCOMES:
Health of the Nation Outcome Scales (HoNOS) | Change from baseline (T0) to 24 months (T3)
  The HoNOS will be used to assess changes in participant's functioning. It will be rated by key worker on a 5-point Likert scale in terms of the following items: 1) aggression, 2) self-harm, 3) substance use, 4) cognitive dysfunction, 5) physical disability, 6) hallucinations and delusions, 7) depression, 8) other symptoms, 9) personal relationships, 10) overall functioning, 11) residential problems, 12) occupational problems. The summed-up total-score ranges from 0 to 48 with lower score indicating better functioning.
Global Assessment of Functioning (GAF) | Change from baseline (T0) to 24 months (T3)
  The GAF is a scale rated by key worker and will be used to assess changes in participant's functioning. Illness severity is rated as a single item based on psychopathology and functioning on a 1 to 100 scale with higher score as indicator for better functioning.
Manchester Short Assessment of Quality of Life (MANSA) | Change from baseline (T0) to 24 months (T3)
  The MANSA is an interview and will be used to assess changes in participant's quality of life. It consists of three sections with total 25 items: 1) personal details, consistent over time (date of birth, gender, diagnosis), 2) personal details, potentially varying over time and to be redocumented if change has occurred (education, employment, income, state benefits, living situation, people the participant lives with, type of residence), and 3) 16 questions that are asked every time. Four of the section three questions are termed objective and are to be answered with yes/no. Twelve of the section three questions are called subjective and ask for answering participant's satisfaction on a 7-point Likert scale. The final score will be computed by averaging the 12 individual items with higher score indicates higher quality of life.
Symptom Check List (SCL-K-9) | Change from baseline (T0) to 24 months (T3)
  The SCL-K-9 is a questionnaire and will be used to assess changes in participant's mental state on a 5-point Likert scale, including items from all of the nine subscales of the original SCL-90-R: 1) depression, 2) anxiety, 3) somatization, 4) phobic fear, 5) obsessive-compulsive, 6) psychoticism, 7) social insecurity, 8) paranoid thinking, 9) hostility. The total-score ranges from 0 to 36 with lower score indicating better mental states.
Diagnoses according to International Classification of Diseases 10 (ICD-10 diagnoses) | The diagnoses will be assessed at baseline (T0) and after 24 months (T3)
  Clinical records
Camberwell Assessment of Need Short Appraisal Schedule (CANSAS) | Change from baseline (T0) to 24 months (T3)
  The CANSAS is an interview and will be used to assess changes in participant's needs in 22 health and social domains on a 3-point Likert scale (no problem; met need; unmet need). For interpretation, the met and unmet needs each will be summed-up.
Oxford Capabilities Questionnaire - Mental Health (OxCAP) | Change from baseline (T0) to 24 months (T3)
  The OxCAP is a questionnaire and will be used to assess changes in participant's capabilities that covers the following domains of functioning and welfare based on 16 items to answer on a 5-point Likert scale: 1) life, 2) bodily health, 3) bodily integrity, 4) senses, imagination and thought, 5) emotions, 6) practical reason, 7) affiliation, 8) species, 9) play, and 10) control over one's environment. The initial index total-score ranges from 16 to 80 and is converted into a standardised 0 to 100 final score with higher score indicating better capabilities.
Important life events, measured with a single item | Important life events will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  Important Life Events for the last six months (at baseline) or since the last assessment, respectively. Free text with subsequent coding
Social Support | Change from baseline (T0) to 24 months (T3)
  A self-generated questionnaire will be used to measure changes in participant's social and living support. The questionnaire consists of 24 items to be answered on a 5-point Likert scale. Total score rages from 24 to 120 with higher score indicating higher support.

OTHER OUTCOMES:
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 1 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The first question records the participants' main source of income: Salary, pension, social benefits, family support, other. No score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 2 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The second question asks for the net income in Swiss Francs.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 3 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The third question asks the whereabouts in recent six months (own apartment, with partner, with family, being homeless, other). No score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 4 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The fourth question asks for any health care utilization for physical health problems (inpatient/outpatient). The format for each answer is 1/0. No score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 5 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The fifth question asks for any health care utilization for mental health problems (inpatient/outpatient). The format for each answer is 1/0. No total or mean score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 6 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The sixth question asks for any intake of psychotropic medication. No score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 7 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The seventh question asks for any contact with the criminal justice services. No score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 8 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The eighth question asks for any internet access. No score will be calculated.
Client Sociodemographic and Service Receipt Inventory - adapted (CSSRI-EU); Question 9 | The CSSRI-EU will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  The CSSRI-EU is an interview and will be used to assess participant's specific sociodemographic details and service utilization. The ninth question asks for any other support utilized in the past six months (daycare, workshops, vocational rehabilitation, integration services, self-help groups, other). No score will be calculated.
Mean number and duration of contacts with service user in IHS | Contact frequency and duration will be assessed at baseline (T0), after 6 months (T1), 12 months (T2), and after 24 months (T3)
  Activity recording with medical tariff (TARMED) reimbursement tool
Independent Housing and Support for people with mental disorders - Fidelity Scale [Selbstbestimmtes Wohnen mit Unterstützung für Menschen mit psychischen Beeinträchtigungen - Modelltreue Skala (SeWo-Psych)] | Model Fidelity will be assessed in months 1-3 and again in month 45.
  The SeWo-Psych is an interview and will be used to assess model fidelity of the residential rehabilitation service Independent Housing and Support (IHS) to be conducted with heads of rehabilitation services. The 32 items are to be answered on a 5-point Likert scale, with higher score indicating higher fidelity. Score will be summed up to a total-score.
Housing First Fidelity Scale | Comparability to HF-Programs will be assessed in months 1-3 and again in month 45.
  The Housing First Fidelity Scale is a 38-item interview assessing model fidelity in Housing First (HF) Programs asking for the following subscales on a 5-point Likert scale: 1) housing choice and structure, 2) separation of housing and clinical services, 3) service philosophy, 4) service array, and 5) program structure. It will be assessed to enhance comparability of IHS in Switzerland with HF-Programs. Items were answered by heads of each rehabilitation service on a 5-point Likert scale, with higher score representing higher similarity with HF-Programs.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Richter, PhD, Principal Investigator — Bern University Hospital for Mental Health
Locations (2):
- Switzerland (2):
  - University Hospital for Mental Health Bern, Center for Psychiatric Rehabilitation, Bern
  - Psychiatric University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richter D, Hoffmann H. Independent housing and support for people with severe mental illness: systematic review. Acta Psychiatr Scand. 2017 Sep;136(3):269-279. doi: 10.1111/acps.12765. Epub 2017 Jun 16. PMID 28620944
- [Background] Richter D, Hoffmann H. Preference for Independent Housing of Persons with Mental Disorders: Systematic Review and Meta-analysis. Adm Policy Ment Health. 2017 Nov;44(6):817-823. doi: 10.1007/s10488-017-0791-4. PMID 28160182
- [Derived] Adamus C, Motteli S, Jager M, Richter D. Independent Supported Housing vs institutional housing rehabilitation settings for non-homeless individuals with severe mental illness - longitudinal results from an observational study. BMC Psychiatry. 2024 Aug 9;24(1):554. doi: 10.1186/s12888-024-05995-7. PMID 39123200
- [Derived] Adamus C, Motteli S, Jager M, Richter D. Independent Supported Housing for non-homeless individuals with severe mental illness: Comparison of two effectiveness studies using a randomised controlled and an observational study design. Front Psychiatry. 2022 Nov 10;13:1033328. doi: 10.3389/fpsyt.2022.1033328. eCollection 2022. PMID 36440393
- [Derived] Motteli S, Adamus C, Deb T, Frobel R, Siemerkus J, Richter D, Jager M. Independent Supported Housing for Non-homeless People With Serious Mental Illness: A Pragmatic Randomized Controlled Trial. Front Psychiatry. 2022 Jan 21;12:798275. doi: 10.3389/fpsyt.2021.798275. eCollection 2021. PMID 35126208
- [Derived] Adamus C, Motteli S, Jager M, Richter D. Independent Housing and Support for non-homeless individuals with severe mental illness: randomised controlled trial vs. observational study - study protocol. BMC Psychiatry. 2020 Jun 19;20(1):319. doi: 10.1186/s12888-020-02712-y. PMID 32560681